CLINICAL TRIAL: NCT03093220
Title: Molecular Typing of Adult Community-acquired Pneumonia in China
Brief Title: Molecular Typing of Community-acquired Pneumonia Based on Multiple-omic Data Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: CapitalBio Group Corporation (Unknown); Chinese Academy of Sciences (Other Government); West China Hospital (Other); Second Hospital of Jilin University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Other Study IDs: 2016YFC0903800
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Infections; Genetic Disorder; Community-Acquired Infections; Host-Pathogen Interactions
MeSH Terms: conditions — Respiratory Tract Infections; Genetic Diseases, Inborn; Community-Acquired Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Lower respiratory tract specimens including sputum, endotracheal aspiration and bronchoalveolar lavage fluid.
  2. Peripheral whole blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- community-acquired pneumonia: all adult patients (aged > 16 years) admit to the 4 hospitals between March 2017 and March 2018 with CAP will be enrolled

SUMMARY:
Community-acquired pneumonia (CAP) is a heterogeneous disease causing great morbidity, mortality and health care burden globally. Typing methods for discriminating different clinical conditions of the same disease are essential to a better management of CAP. Traditional typing systems based separately on clinical manifestations (such as PSI and CURB-65), pathogens(bacterial types, virulence, drug resistance, etc) or host immune state (immunocompetent, immunocompromised or immunodeficiency). Thus, they are barely able to represent the real disease status nor to precisely predict the mortality.

As the development of multi-omic technologies, the relatedness of different phenotypes at a molecular level have revolutionized our ability to differentiate among patients. Our study is aimed at establishing a novel molecular typing method of CAP. Multi-omic (including genomics, transcriptomes, and metabolisms) data obtained from enrolled CAP patients and isolated pathogens would be integrated analyzed and interpreted. Tthe investigators believe that an appropriate molecular typing method would lead to revolutionary changes in current arrangements of CAP.

ELIGIBILITY:
Inclusion Criteria:

* adult (aged > 16 years)
* diagnosed as community-acquired pneumonia

Exclusion Criteria:

* being immunocompromised, including history of glucocorticoid taken for more than 1 month, history of immunosuppressive therapy, history of human immunodeficiency virus (HIV) infection, solid tumor or hematological malignancy
* history of long-term nursing home stays
* history of recently hospitalized (<90 days)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all adult patients (aged > 16 years) admit to the 4 hospitals between March 2017 and March 2018 with CAP
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
30 day mortality | 30 days after the onset of CAP
  all-cause death in 30 days after the onset of CAP

SECONDARY OUTCOMES:
complications | 30 days after the onset of CAP
  nonfatal complications including critical organic or systematic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Zhancheng Gao, Professor, Study Chair — Department of Respiratory Critical Care Medicine
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen L, Xue J, Zhao L, He Y, Fu S, Ma X, Yu W, Tang Y, Wang Y, Gao Z. Lysophosphatidylcholine acyltransferase level predicts the severity and prognosis of patients with community-acquired pneumonia: a prospective multicenter study. Front Immunol. 2024 Jan 8;14:1295353. doi: 10.3389/fimmu.2023.1295353. eCollection 2023. PMID 38259459
- [Derived] Yin L, Zhang Y, Zheng Y, Luo Q, Zhao L, Ni W, Xu Y, Gao Z. Early Detection of Aspergillus Species in Lower Respiratory Tract is Associated with Higher Mortality in Viral Community-Acquired Pneumonia: A Multicenter Prospective Cohort Study in China. Lung. 2023 Aug;201(4):387-396. doi: 10.1007/s00408-023-00638-2. Epub 2023 Jul 22. PMID 37480410
- [Derived] Xie Y, Yu Y, Zhao L, Ning P, Luo Q, Zhang Y, Yin L, Zheng Y, Gao Z. Specific Cytokine Profiles Predict the Severity of Influenza A Pneumonia: A Prospectively Multicenter Pilot Study. Biomed Res Int. 2021 Oct 13;2021:9533044. doi: 10.1155/2021/9533044. eCollection 2021. PMID 34692846
- [Derived] Chen L, Zhao L, Shang Y, Xu Y, Gao Z. Admission lysophosphatidylethanolamine acyltransferase level predicts the severity and prognosis of community-acquired pneumonia. Infection. 2021 Oct;49(5):877-888. doi: 10.1007/s15010-021-01585-x. Epub 2021 Mar 10. PMID 33694084
- [Derived] Zheng Y, Ning P, Luo Q, He Y, Yu X, Liu X, Chen Y, Wang X, Kang Y, Gao Z. Inflammatory responses relate to distinct bronchoalveolar lavage lipidome in community-acquired pneumonia patients: a pilot study. Respir Res. 2019 May 2;20(1):82. doi: 10.1186/s12931-019-1028-8. PMID 31046764
- [Derived] Luo Q, He X, Ning P, Zheng Y, Yang D, Xu Y, Shang Y, Gao Z. Admission Pentraxin-3 Level Predicts Severity of Community-Acquired Pneumonia Independently of Etiology. Proteomics Clin Appl. 2019 Jul;13(4):e1800117. doi: 10.1002/prca.201800117. Epub 2019 Feb 12. PMID 30557448
- [Derived] Ning P, Zheng Y, Luo Q, Liu X, Kang Y, Zhang Y, Zhang R, Xu Y, Yang D, Xi W, Wang K, Chen Y, An S, Gao Z. Metabolic profiles in community-acquired pneumonia: developing assessment tools for disease severity. Crit Care. 2018 May 14;22(1):130. doi: 10.1186/s13054-018-2049-2. PMID 29759075
- [Derived] Luo Q, Ning P, Zheng Y, Shang Y, Zhou B, Gao Z. Serum suPAR and syndecan-4 levels predict severity of community-acquired pneumonia: a prospective, multi-centre study. Crit Care. 2018 Jan 24;22(1):15. doi: 10.1186/s13054-018-1943-y. PMID 29368632